CLINICAL TRIAL: NCT05451706
Title: Improving College Students' Mental Help-Seeking Intention During the COVID-19 Pandemic
Acronym: MHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Qiwei Luna Wu, Assistant Professor, Cleveland State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ClevelandSU
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Help-Seeking Behavior; Mental Health Issue
Keywords: Mental help-seeking; COVID-19; College students; Self-persuasion
MeSH Terms: conditions — Help-Seeking Behavior; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YouTube Intervention (Experimental): Participants assigned to this task were asked to search YouTube for a 5-10 minutes' video promoting mental help-seeking among college students. Then, they were expected to provide the link to the video and describe the content of the video. Next, participants were guided to form rebuttals disapproving three statements that rationalize students' low intention to seek mental help.
  Interventions: Behavioral: Mental help-seeking self-persuasion
- Facebook Intervention (Active Comparator): This task was to draft a Facebook message for the participants' fellow students. In their message, participants were expected to list three reasons for seeking mental help. The length of the message was not pre-determined.
  Interventions: Behavioral: Mental help-seeking self-persuasion
- YouTube Control Group (Placebo Comparator): Participants in this group were assigned a YouTube task advocating social distancing during a pandemic. The question prompts were modified from the tasks for the experimental groups.
  Interventions: Behavioral: Mental help-seeking self-persuasion
- Facebook Control Group (Placebo Comparator): Participants in this group were assigned a Facebook task advocating social distancing during a pandemic. The question prompts were modified from the tasks for the experimental groups.
  Interventions: Behavioral: Mental help-seeking self-persuasion

INTERVENTIONS:
Behavioral: Mental help-seeking self-persuasion — Employing a longitudinal design, this study used a self-persuasion framework in a 4-arm intervention to increase college students' help-seeking intentions during the COVID-19 pandemic.

SUMMARY:
This study aimed at testing the effectiveness of a longitudinal intervention in increasing college students' intention to seek mental help during the pandemic.

DETAILED DESCRIPTION:
This study aimed at testing the effectiveness of a longitudinal intervention in increasing college students' intention to seek mental help during the pandemic.

A four-armed randomized controlled experiment was conducted to compare two self-persuasion methods against two control conditions. Assessments took place at baseline (T0), post-first treatment (T1), post-second treatment (six weeks, T2), and ten-week follow-up (T3).

The results showed that the intervention significantly increased students' help-seeking intention, attitude, and efficacy at different time points. It also reduced mental help-seeking-related stigma after the first task.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Full-time undergraduate students
* Had more than a moderate amount of mental distress

Exclusion Criteria:

* Under 18 years old
* Not full-time undergraduate students
* Had less than a moderate amount of mental distress

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 926 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Help-Seeking Intention | 10 weeks
  Help-Seeking Intention was measured by one item created based on recommendations by Ajzen (2002). Measured on a 5-point scale (1 = extremely unlikely, 5 = extremely likely), this item asked, "If you have a personal-emotional problem, how likely is it that you would seek help from a mental health professional (a psychologist, psychologist, or psychotherapist)?" Higher scores on this item suggest higher intentions to seek professional mental help.
Help-Seeking Behavior | 10 weeks
  Help-Seeking Behavior was measured by a validated item modified from previous research based on the transtheoretical model (Sarkin et al., 2001). The item asked about if a participant has sought mental help from a health care professional. Answers to this item included "1 = not intending to seek help in the next six months," "2 = intending to seek help in the next six months," "3 = planning to seek help in the next 30 days," "4 = have already sought help but for less than six months," and "5 = have been under treatment for more than six months."

SECONDARY OUTCOMES:
Mental help-seeking attitudes | 10 weeks
  participants rated 1 ("strongly disagree") to 5 ("strongly agree") on ten items of the Attitudes Toward Seeking Professional Psychological Help Scale-Short Form (ATSPPHS-SF) (Fischer & Farina, 1995).
Self-stigma of seeking mental help | 10/2020 - 1/10 weeks
  Participants rated 1 ("strongly disagree") to 5 ("strongly agree") on ten items adopted from the Self-Stigma of Seeking Help (SSOSH) scale (Vogel et al., 2006).
Mental help-seeking efficacy | 10 weeks
  Mental Help-Seeking Efficacy was measured by five items modified from previous research (Mo & Mak, 2009) and recommendations (Ajzen, 2002). Participants rated 1 ("strongly disagree") to 5 ("strongly agree") on the answers.

CONTACTS AND LOCATIONS:
Overall Officials: Qiwei Wu, Principal Investigator — Cleveland State University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as required by the IRB protocol.